CLINICAL TRIAL: NCT05857540
Title: The Effects of Upper-Extremity Plyometric Combined Strength Training in Overhead Athletes With Shoulder Instability
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM111161F
Record Dates: First submitted 2023-04-11; First posted 2023-05-12 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Glenohumeral Subluxation; Shoulder Subluxation; Shoulder Instability Subluxation Bilateral
Keywords: Plyometric; Strengthening; Overhead athlete; Shoulder instability
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plyometric training group (Experimental): Participants in this group will receive upper extremity plyometric training in body weight or with weight ball and strengthening exercises with band, dumbbell and barbell. The difficulty and intensity of the movement protocol will increase weekly. They will be trained 2 times per week for 6 weeks with an average duration of 50 min per session.
  Interventions: Procedure: Plyometric and strengthening exercises
- Strengthening training group (Active Comparator): Participants in this group will receive upper extremity strengthening exercises with band, dumbbell and barbell. The intensity of the movement protocol will increase weekly. They will be trained 2 times per week for 6 weeks with an average duration of 50 min per session.
  Interventions: Procedure: Strengthening exercise

INTERVENTIONS:
Procedure: Plyometric and strengthening exercises — Each session includes 2 upper-extremity plyometric exercises in bodyweight or with weight ball for 15-20 minutes and 4-5 strengthening exercises with band, dumbbell or barbell for 30-35 minutes. The difficulty of the movement protocol will increase weekly. They will be trained 2 times per week for 6 weeks with an average duration of 50 min per session.
  Arms: Plyometric training group
Procedure: Strengthening exercise — Each session includes 5 upper-extremity strengthening exercises with band, dumbbell or barbell for 50 minutes. The difficulty of the movement protocol will increase weekly. They will be trained 2 times per week for 6 weeks with an average duration of 50 min per session.
  Arms: Strengthening training group

SUMMARY:
The purpose of this randomized controlled trial is to investigate the additional effects of upper extremity plyometric training versus strength training alone in recreational overhead athletes with shoulder instability. The investigators hypothesis that compared to strengthening training alone, plyometric training combined with strengthening training will significantly improve shoulder isokinetic strength, proprioception, scapular kinematics, symptoms of shoulder instability, and shoulder function.

DETAILED DESCRIPTION:
Background: Shoulder instability is a common problem in active young adults with a wide spectrum ranging from microinstability, subluxation to dislocation. In patients with instability of Stanmore polar type 2 or 3, recurrent shoulder instability may be related to abnormal movement patterns but not result from trauma. Non-operative management is suggested to this subgroup as the first-line treatment. Previous rehabilitation protocols including progressive shoulder muscles strengthening and neuromuscular control training have shown positive effects on functional outcomes in individuals with shoulder instability. Recent protocols for shoulder instability usually include various types of plyometric training to prepare injured athletes to return to sports. Plyometric training in lower extremity has been wildly used for knee injury prevention. In upper extremity, plyometrics also has been shown to improve isokinetic strength, throwing performance, and proprioception in healthy subjects and healthy overhead athletes. However, it is still not well-understood that whether a strengthening training combined with plyometrics would be more effective to improve shoulder neuromuscular control and shoulder function in subjects with instability. The purpose of this study is to investigate the additional effects of upper extremity plyometric training in recreational overhead athletes with anterior shoulder instability. The investigators hypothesis that compared to strengthening training alone, plyometric training combined with strengthening training will significantly improve strength, proprioception, shoulder kinematic and muscle activity, shoulder pain and shoulder function.

Methods: A total of 64 participants with anterior shoulder instability will be randomized to either an experimental group (plyometric and strengthening training) or a control group (strengthening training). Both groups will receive a 50-minute supervised training protocol twice a week for 6 weeks. The primary outcomes include (1) isokinetic assessment of internal and external rotation (peak torque, time to peak torque, and amortization time); (2) proprioception (active and passive joint position sense); (3) seated medicine ball throw test (distance in cm). The secondary outcomes include (1) shoulder pain and instability with 10-cm visual analogue scale (VAS); (2) shoulder function assessed with the Disability of Arm, Shoulder and Hand (DASH) questionnaire; (3) Global rating of change (GRC). GRC will be measured after the end of 12 session of intervention, and all the other outcomes will be measured at baseline and following 12 sessions of exercise training. The two-way repeated measures ANOVAs will be used to compare primary and secondary outcome variables between groups. The significant level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Have experience of at least 1 of the following symptoms of shoulder instability during upper extremity movement: (a) pain, clicking, a sense of the shoulder coming apart, (b) dead-arm syndrome, or (c) subluxation of the joint.
2. Self-reported decreased performance or feeling fear to perform shoulder movements during sports or daily activities
3. Positive findings on ≥ 1 of the following 5 tests: load and shift test, apprehension, relocation, & surprise tests, Gagey hyperabduction test, sulcus sign, Feagin test
4. Recreational overhead athletes who keep practicing ≥ 4 hours/week in the recent 1 month and with ≥ 1 year overhead sports experience

Exclusion Criteria:

1. Full contact sport athletes
2. Severe shoulder instability with > 5 shoulder dislocations history
3. Obvious shoulder bony/labrum lesion in the dominant side warranted for surgery first as decided by the orthopedic surgeon
4. Previous surgery or fracture in the shoulder area on the dominant side within 1 year
5. Voluntary instability (the ability to deliberately dislocate one's shoulder)
6. During acute phase after shoulder dislocation event
7. Not suitable to start plyometric training yet: Shoulder muscle weakness (manual muscle test <3) or range of motion limitation (<90 abduction, <70 external rotation) in the dominant side
8. Pregnancy
9. Cancer, neck pain, brain & neurological impairment
10. Ehlers-Danlos syndrome or Marfan syndrome
11. Unable to attend 6 weeks supervised training

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder isokinetic muscle strength | Change from baseline shoulder isokinetic muscle strength through completion of 12-session intervention, an average of 6 weeks
  Shoulder isokinetic muscle strength will be measured by dynamometer in 3 modes (concentric/concentric, concentric/eccentric, eccentric/concentric) at 3 angular velocities (90°/s, 180°/s, & 240°/s), 1 set of 5 repetitions for each angular velocities. Shoulder isokinetic muscle strength will be normalized by body weight (BW) and described with peak torque/BW (N·m·kg-1).
Shoulder acceleration time, deceleration time, and amortization time | Change from baseline shoulder isokinetic muscle strength through completion of 12-session intervention, an average of 6 weeks
  Shoulder acceleration time, deceleration time, and amortization time will be measured by dynamometer in concentric/concentric mode at 3 angular velocities (90°/s, 180°/s, & 240°/s) and will be described with millisecond (ms).
Shoulder proprioception | Change from baseline shoulder external rotation joint position sense through completion of 12-session intervention, an average of 6 weeks
  Shoulder proprioception will be measured by dynamometer in 90° shoulder abduction and 90° elbow flexion position, including active joint position sense and passive joint position sense. The proprioception will be described with degree of error from target position.
Seated medicine ball throw distance | Change from baseline seated medicine ball throw distance through completion of 12-session intervention, an average of 6 weeks
  Subjects will throw a 2kg soft weighted ball as far forward as possible with dominant arms while sitting with back against a wall and legs bending with feet flat on the floor. Outcomes include average throwing distance and maximal throwing distance (cm). The distances are measured with measure tape.

SECONDARY OUTCOMES:
Shoulder function | Change from baseline DASH questionnaire through completion of 12-session intervention, an average of 6 weeks
  Shoulder function will be measured by the disabilities of the arm, shoulder and hand (DASH) questionnaire, including the disability/symptom section (30 items, scored 1-5) and the optional high performance Sport/Music or Work section (4 items, scored 1-5). A higher score indicates greater disability.
Visual analogue scale (VAS) of shoulder pain and instability | Change from baseline VAS of shoulder pain and instability through completion of 12-session intervention, an average of 6 weeks
  Shoulder pain and instability will be measured by visual analogue scale (VAS). Subjects need to mark the point that they feel represent their perception of their current state on a 10-cm line. Scores range from 0 (no symptom) to 100 (maximum symptom).
Global rating of change (GRC) | through completion of 12-session intervention, an average of 6 weeks
  The improvements in a patient's condition will be measured with 15-point self-report GRC scale. Score ranges from -7 (lack of progress) to 7 (maximum of progress).

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taipei, Taiwan